CLINICAL TRIAL: NCT00728000
Title: Phase II Study Of Neoadjuvant Chemotherapy With Gemcitabine, Oxaliplatin And Erlotinib (Gemoxt) In Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Phase II Study Of Neoadjuvant Chemotherapy In Borderline Resectable Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study withdrawn due to lack of enrollment
Sponsor: University of Cincinnati (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-06-030; OX-06-030
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy regimen (Experimental): Gemcitabine and oxaliplatin are given intravenously (into the vein) every 2 weeks. Erlotinib is a pill that is taken by mouth daily.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Erlotinib

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2 IV on day 1 and day 15 over 30mins.
  Other Names: Gemzar®
Drug: Oxaliplatin — 100mg/m2 IV on days 1 and 15 given over 120 mins.
  Other Names: Eloxatin
Drug: Erlotinib — 100mg/day PO on days 1-14 and 15-28
  Other Names: Tarceva

SUMMARY:
The goal of this study is to determine the effect of chemotherapy on decreasing the size of unresectable pancreas cancer thereby allowing it to be surgically removed. In addition, this study may provide information on how tumors behave when exposed to certain types of chemotherapy.

DETAILED DESCRIPTION:
Although surgery is the only curative modality for pancreatic adenocarcinoma, the majority of patients (~80%)are unresectable at presentation. The use of a multimodality approach may be a crucial method to improve the dismal survival rate of patients with pancreatic cancer. A logical tactic is to use neoadjuvant cytotoxic agents and targeted drugs to facilitate resectability.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic or cytologic diagnosis of pancreatic adenocarcinoma. Patients with endocrine tumors or lymphoma of the pancreas are ineligible.
* Patients must have locally advanced disease that is considered to be "borderline" surgically resectable (see Section 4.0). Patients with metastatic disease or grossly resectable disease on presentation are ineligible.
* Patients must have measurable disease prior to starting this study. Patients with primarily non-measurable disease, including lesions to small to be characterized, effusions, ascites, diffuse bone disease, diffuse skin disease, leptomeningeal disease, lymphangitis, pneumonitis or disease measured by indirect or biochemical means, are not eligible. Testing for measurable disease must have been completed 28 days prior to registration.
* Patients must consent to utilization of tissue for research in this protocol. Tissue will be evaluated via immunohistochemical staining for deoxycytidine kinase, ERCC-1 and ERCC-2 (XPD). Patients may be asked if they are willing to allow their tissue to be used for future studies that are not defined in this protocol. Disallowing the use of tissue for future studies does not limit eligibility in this protocol.
* Patients must fulfill the required initial laboratory data to be obtained within 28 days prior to registration: AGC ≥ 1,500cells/μL, Platelet ≥ 100,000cells/μL, Hgb > 8.0 g/dl, Bilirubin ≤ 2.0 X IULN, Serum Creatinine ≤ 2.0mg/dL, AST(SGOT) ≤ 2.5x IULN, ALT(SGPT) ≤ 2.5x IULN, CA19-9 (any value),
* Patients must have an ECOG/Zubrod performance status of 0-2.
* Patients must be able to read and understand English in order to participate in this study, or have a certified translator present.
* Due to the potentially harmful effects of chemotherapy on a developing fetus, patients who are pregnant are planning to become pregnant, or who are lactating should not participate in this study.
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* All patients must be informed of the investigational nature of this study and must sign, date and give written consent in accordance with institutional and federal guidelines.
* All patients must be18 years of age or older to participate.

Exclusion Criteria:

* Patients with known brain metastases are ineligible. Brain imaging studies are not required for eligible patients with no neurologic signs or symptoms. If brain imaging studies are performed, they must be negative for disease.
* Patients who have had prior surgery for their pancreatic carcinoma are not eligible for this study. This does not include patients who have had cytologic brushing, fine needle aspiration or core biopsy of their tumor for diagnostic purposes.
* Patients must not have received prior chemotherapy, radiotherapy, chemoradiotherapy, surgery, immunotherapy or hormonal therapy for pancreatic cancer.
* Patients must not have received prior erlotinib or other therapies that target EGFR. Patients must not have received prior tyrosine kinase inhibitors.
* Have a significant history of uncontrolled cardiac disease including uncontrolled hypertension, unstable angina or uncontrolled congestive heart failure.
* Have a significant history of intersitital lung disease
* Have a significant history of peripheral neuropathy (grade must be <1) or mononeuropathy multiplex.
* Have temperature >101.30 F or active infection
* No other history of malignancy is allowed except for the following:

adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.

* There must be no other plans for the patient to receive concurrent chemotherapy, radiotherapy, chemoradiotherapy, surgery, immunotherapy or hormonal therapy for the treatment of their cancer while on protocol.
* Due to the undetermined effect of chemotherapy in patients with HIV infection and the potential for serious interaction with anti-HIV medications, patients who are known to be infected with HIV are not eligible for this study. An HIV test is not required to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is a dichotomous variable evaluating the # of patients who obtain an RO resection versus the number of patients that do not obtain an RO resection plus the number of patients who are not resectable. | 9-10 months

SECONDARY OUTCOMES:
DFS, PFS, OS and TD will be observed on each patient and censored at the end of the study. Measurements of toxicity are categorical variables. All numerical variables will be summarized by mean +- standard deviation (STD) and/or median (range) | 9-10 months

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Oleksowicz, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States